CLINICAL TRIAL: NCT02656329
Title: AdreView™ Myocardial Imaging for Risk Evaluation - A Multicentre Trial to Guide ICD Implantation in NYHA Class II & III Heart Failure Patients With 25%≤LVEF≤35%
Brief Title: International Study to Determine if AdreView Heart Function Scan Can be Used to Identify Patients With Mild or Moderate Heart Failure (HF) That Benefit From Implanted Medical Device
Acronym: ADMIRE-ICD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor discretion (low recruitment rate)
Sponsor: GE Healthcare (Industry)
Collaborators: Advanced Clinical, LLC (Unknown); TFS (Unknown); H2O Clinical LLC (Industry); AG Mednet Inc. (Unknown); ICON CEAC (Unknown); ICON Clinical (Unknown); ABX CRO (Other); TransPerfect (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GE-122-020; 2015-001464-19 (EudraCT Number)
Record Dates: First submitted 2016-01-07; First posted 2016-01-14 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
Keywords: Heart Failure (HF); Single photon emission computer tomography scan (SPECT); Implantable cardioverter defibrillator (ICD); Left Ventricular ejection fraction (LVEF); New York Health Association (NYHA); Metaiodobenzylguanidine (mIBG); 123I-iobenguane; Heart-to-mediastinal ratio (H/M); ADMIRE-ICD (AdreView Myocardial Imaging for Risk Evaluation - Implantable Cardioverter Defibrillator; All-cause mortality; Cardiac mortality
MeSH Terms: conditions — Heart Failure | interventions — 3-Iodobenzylguanidine; Defibrillators, Implantable; thyroid stimulation-blocking antibody; Potassium Iodide; potassium perchlorate; Lugol's solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AdreView™ (Experimental): Participants received 1 intravenous injection of 10 mCi (370 MBq) of AdreView™ (Iobenguane I-123 Injection). Participants with AdreView™ Heart-to-Mediastinal ratio (H/M) <1.6 underwent Implantable Cardioverter Defibrillator (ICD) device implantation and H/M >= 1.6 continued to receive Guideline-Directed Optimal Medical Therapy (GDMT) according to clinical standard practice.
  Interventions: Drug: Iobenguane I -123 Injection; Device: Implantable Cardioverter Defibrillator; Drug: Thyroid blocking
- Standard of Care (Experimental): Participants received 1 intravenous injection of 10 mCi (370 MBq) of AdreView™ (Iobenguane I-123 Injection) and underwent ICD implantation and were followed up in accordance with internationally accepted Heart Failure (HF) guidelines.
  Interventions: Drug: Iobenguane I -123 Injection; Device: Implantable Cardioverter Defibrillator

INTERVENTIONS:
Drug: Iobenguane I -123 Injection — Iobenguane I-123 Injection, AdreView. All participants scheduled for an Iobenguane I-123 Injection, AdreView scan.
  Other Names: AdreView; Iobenguane I-123 Injection
  Arms: AdreView™
Device: Implantable Cardioverter Defibrillator — In the Iobenguane I-123 Injection group, participants with H/M ratio less or equal to 1.6 underwent ICD device implantation, while those with H/M ratio greater than or equal to 1.6 did not undergo ICD implantation.
  Arms: AdreView™
Drug: Thyroid blocking — Participants received a thyroid blocking agent before the Iobenguane I-123 Injection, AdreView, scan unless medically not indicated, according to local practice.
  Other Names: Potassium Iodide; Potassium Perchlorate; Lugol's Solution
  Arms: AdreView™
Drug: Iobenguane I -123 Injection — Iobenguane I-123 Injection, AdreView. All participants scheduled for an Iobenguane I-123 Injection, AdreView scan.
  Other Names: AdreView; Iobenguane I-123 Injection
  Arms: Standard of Care
Device: Implantable Cardioverter Defibrillator — All participants allocated to the SoC (control) group underwent ICD implantation.
  Arms: Standard of Care

SUMMARY:
This is an event-driven Phase IIIb, multicentre, randomised, clinical study to demonstrate the efficacy of AdreView™ imaging for appropriately guiding the decision of implantable cardioverter defibrillator (ICD) implantation, in New York Health Association (NYHA) class II and III heart failure participants with 25%<=left ventricular ejection fraction (LVEF)<=35%, and in particular, for identifying participants who are at low risk for sudden cardiac death and who would not benefit, or may suffer harm, from implantation of an ICD device.

ELIGIBILITY:
Inclusion Criteria:

* Participants >=18 years of age at the time dated informed consent was obtained.
* Female participants must be pre-menarchal, surgically sterile (had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (cessation of menses for more than 1 year), non-lactating, or, if of childbearing potential, a serum or urine pregnancy test with the results known prior to AdreView (Iobenguane I-123 Injection) administration) was negative.
* Participants willing and able to comply with all study procedures and a signed and dated informed consent was obtained before any study-procedure was carried out.
* Heart failure NYHA class II or III for symptoms, participants with ischemic or non-ischemic heart disease, eligible for ICD implantation as per each site's standard of practice.
* Non-ischemic dilated cardiomyopathy or ischemic heart disease of at least 3 months duration receiving guideline-directed optimal medical therapy.
* 25%≤LVEF≤35%, performed within 3 months before or at time of enrollment, as measured by radionuclide ventriculography, or electrocardiogram [ECG]-gated SPECT myocardial perfusion imaging [MPI], or magnetic resonance imaging [MR], computed tomography [CT], or 3D or 2D echocardiography [Simpson's or multidisc method only, M-mode echocardiography was not accepted].

In case LVEF measurement was performed within 3 months before enrollment, measurement should be performed at least 40 days after a hospitalization for HF or acute coronary syndrome (including myocardial infarction), and to be valid, method of measurement should be in accordance with the protocol and the imaging exam should be made available to the Sponsor in digital format. In case several valid LVEF measurements are available, the closest to enrollment will be used for inclusion determination.

* Clinically stable heart failure in the medical judgment of the investigator (i.e. no significant changes in medication, no worsening of symptoms, no unscheduled visits to the doctor's office) for the past 30 days and no hospitalization for heart failure or acute coronary syndrome (including myocardial infarction) in the past 40 days.
* Reasonable expectation of meaningful survival for at least 1 year.

Exclusion Criteria:

* Participants with existing ICD or participant having an indication of ICD implantation for secondary prevention of sudden cardiac death.
* Hospitalization for HF or for acute coronary syndrome in the previous 40 days.
* Participants where a cardiac resynchronisation therapy (CRT) was planned or indicated.
* Other indication for placement of device (sustained ventricular tachycardia, resuscitated sudden death, need for atrioventricular pacing).
* NYHA class I or class IV symptoms at the time of study entry.
* Participants with chronic renal insufficiency defined as serum creatinine ≥ 3 mg/dl (or ≥ 265.2 µmol/L).
* American College of College-American Heart Association (ACC-AHA) class III or class IV (unstable) angina.
* Known or suspected hypersensitivity/allergy to Iobenguane or to any of the excipients an Adreview (Iobenguane I-131 injection).
* Participant who was pregnant or plans to become pregnant within 2 weeks after AdreView (Iobenguane I-123 Injection) administration.
* Participant who had used any medication in the 2 weeks before AdreView (Iobenguane I-123 Injection) that could interfere with the test: e.g. but not limited to amitriptyline or derivatives, imipramine or derivatives, other antidepressants or drugs known or suspected to inhibit the norepinephrine transporter, antihypertensives that deplete norepinephrine stores or inhibit reuptake, sympathomimetic amines or cocaine.
* Participants that had a medical condition that could interfere with the AdreView test (e.g. but not limited to left ventricular assist device (LVAD), or prior heart transplant).
* Participants who participated in a clinical study involving a drug or device within 30 days prior to study entry and participants participating in any other clinical study.
* Participants having serious non-cardiac medical condition associated with significant elevation of plasma catecholamines, including pheochromocytoma.
* Participants with a clinical diagnosis of (or being treated for) Parkinson's disease or Multiple System Atrophy.
* The participant had participated in a research study using ionizing radiation in the previous 12 months.
* Participants previously randomized in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (94):
- United States (29):
  - Vascular Biology and Hypertension Program, University of Alabama at Birmingham, Birmingham, Alabama
  - Comprehensive Cardiovascular Medical Group, Bakersfield, California
  - Sharp Grossmont Hospital, La Mesa, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - VA Connecticut Healthcare System (VACHS), West Haven, Connecticut
  - Cardiology Physicians PA/Red Clay Research, LLC, Newark, Delaware
  - Bethesda Health, Boynton Beach, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Cardiology Consultants, Pensacola, Florida
  - South Miami Heart Specialists, South Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - MMP ME Health Cardiology, Scarborough, Maine
  - MedStar Shah Medical Group, Charlotte Hall, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Department of Cardiology, K-14 (Henry Ford Health System), Detroit, Michigan
  - Regions Hospital and Regions Heart Center Clinic, Saint Paul, Minnesota
  - University at Buffalo, Buffalo, New York
  - Advanced Cardiology Group, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - WakeMed, Raleigh, North Carolina
  - Veterans Affairs North Texas Healthcare System, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Texas Institute of Cardiology, PA, McKinney, Texas
  - Victoria Heart and Vascular Center, Victoria, Texas
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - CIUSSS de L'Estrie - CHUS Hopital Fleurimont, Sherbrooke, Quebec
  - Institut Universitaire De Cardiologie Et De Pneumologie De Quebec, Québec
- Czechia (8):
  - Fakultni nemocnice Brno Bohunice, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - FN Hradec Kralove, Hradec Králové
  - Krajska nemocnice Liberec, Liberec
  - Fakultni nemocnice Plzen, Lochotín
  - Fakultni nemocnice v Kralovske Vinohrady, Prague
  - Fakultni nemocnice v Motole, Prague
  - Masarykova nemocnice v Usti nad Labem, Ústí nad Labem
- France (8):
  - CHR Metz-Thionville - Site de Mercy, Ars-Laquenexy
  - CH Antoine Beclere, Clamart
  - CHU Clermont-Ferrand, 63003 Montalembert, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - CHRU de Lille, Lille
  - Hopital de Rangueil CHU Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
  - Hopitaux de Brabois Chu Nancy, Vandœuvre-lès-Nancy
- Germany (2):
  - Kliniken Maria Hilf GmbH, Klinik fur Nuklearmedizin, Mönchengladbach
  - Klinik & Poliklinik fur Nuklearmedizin, LMU, Campus Grobhader, Munich
- Hungary (7):
  - Varosmajori Sziv es Ergyogyaszati Klinika, Budapest
  - Budai Irgalmasrendi Korhaz, Budapest
  - Gottsegen Gyorgy Orszagos Kardiologiai Intezet, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont Kardiológia Osztály/Nuklearis Medicina Osztaly, Budapest
  - Semmelweis Egyetem Nuklearis Medicina Kozpont, Budapest
  - Debreceni Egyetem, Kardiologia Intezet and ScanoMed Nuclear Medicine Institute, Debrecen
  - Coromed-SMO ft., Pécs
- Italy (10):
  - Azienda Ospedaliera Universitaria G. Martino, Messina
  - Area Cardiologia Critica - IRCCS Centro Cardiologico Mozino, Milan
  - Ospedale Santa Croce, Moncalieri
  - Azienda Ospedaliero-Universitaria Federico II Dipartimento ad Attivita Integrata di Cardiologia,Cardiochirurgia ed Emergenze Cardiovascolari, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carità, Dipartimento Cardiologico, Cardiologia 1, Novara
  - Instituti Clinici Scientifici Maugeri Spa Societa Benefit, Pavia
  - Dipartimento di Scienze Cardiovascolari, Respiratorie Neufrologiche e Geriatriche - Universita di Roma "La Sapienza", Rome
  - Ospedale Santa Maria di Ca' Foncello, Treviso
  - Venezia Mestre - Azienda ULSS 12 "Veneziana", Venezia
  - Ospedale dell'Angelo, 30174, Venezia Mestre, Venice
- Netherlands (5):
  - Onze Lieve Vrouwen Gasthuis, Amsterdam
  - Academic Medical Center, Amsterdam
  - Amphia Zickenhuis, Breda
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
- Poland (7):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny Nr 7 Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Wojskowy Instytut Medyczny, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
  - Dolnośląski Szpital Specjalistyczny im. T. Marciniaka Centrum Medycyny Ratunkowej, Wroclaw
- Spain (11):
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar (Murcia)
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Leon, León
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Son Espases, Palma de Mallorca (Illes Balears)
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Universitario San Juan de Alicante, San Juan Alicante
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela (A Coruña)
  - Hospital General Universitario de Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Study was conducted at 70 centers in United States of America, Canada and Europe between 30 December 2015 and 04 May 2018. A total of 395 participants were enrolled in study, of which 52 were screen failures mainly due to exclusion criteria met.
Pre-assignment Details: Out of 343 participants, 321 participants with 25% <=left ventricular ejection fraction (LVEF) <=35% were randomized in a 1:1 ratio to the AdreView™ group or Standard of Care (SoC) group stratified by enrolling center via an interactive web response system and 22 participants were not randomized but included in safety analysis set.
Groups:
- AdreView™: Participants received 1 intravenous injection of 10 millicurie (mCi) (370 MBq) of AdreView™ (Iobenguane I-123 Injection). Participants with AdreView™ Heart-to-Mediastinal ratio (H/M) <1.6 underwent Implantable Cardioverter Defibrillator (ICD) device implantation and H/M >= 1.6 continued to receive Guideline-Directed Optimal Medical Therapy (GDMT) according to clinical standard practice.
Period: Overall Study
Arm/Group | AdreView™ | Standard of Care
Started | 164 | 157
Completed | 0 | 0
Not Completed | 164 | 157
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Study termination by Sponsor | 150 | 142
Not completed — Other than specified above | 5 | 6

BASELINE CHARACTERISTICS:
Population: Baseline population included randomized participants.
Groups:
- AdreView™: Participants received 1 intravenous injection of 10 mCi (370 MBq) of AdreView™ (Iobenguane I-123 Injection). Participants with AdreView™ Heart-to-Mediastinal ratio (H/M) <1.6 underwent Implantable Cardioverter Defibrillator (ICD) device implantation and H/M >= 1.6 continued to receive GDMT according to clinical standard practice.
- Standard of Care: Participants received 1 intravenous injection of 10 mCi (370 MBq) of AdreView™ (Iobenguane I-123 Injection) and underwent ICD implantation and were followed up in accordance with internationally accepted HF guidelines.
- Total: Total of all reporting groups
Arm/Group | AdreView™ | Standard of Care | Total
Number analyzed (Participants) | 164 | 157 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.40) | 62.1 (10.05) | 63.1 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 22 | 57
  Male | 129 | 135 | 264
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 9 | 26
  Not Hispanic or Latino | 142 | 140 | 282
  Unknown or Not Reported | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 149 | 137 | 286
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: All-cause mortality included all reported deaths of participants during the study due to any cause. Percentage of participants who died due to any cause were reported.
Time Frame: From randomization until the end of the follow-up period (median 304 days)
Population: Analysis was performed on full analysis set (FAS) that was defined as participants included in the safety analysis set who were randomised to the AdreView™ group or the SoC group.
Measure: Number; unit: percentage of participants
Groups:
- AdreView™: Participants received 1 intravenous injection of 10 mCi (370 MBq) of AdreView™ (Iobenguane I-123 Injection). Participants with AdreView™ H/M ratio <1.6 underwent ICD device implantation and H/M ratio >= 1.6 continued to receive GDMT according to clinical standard practice.
Arm/Group | AdreView™ | Standard of Care
Number analyzed (Participants) | 164 | 157
percentage of participants | 3.0 | 3.2
Statistical Analysis 1: Comparison: AdreView™ vs Standard of Care; Analysis was performed using the Cox proportional hazards model stratified by country, with method of treatment guidance (SoC vs AdreView™ group) as the only covariate; Test type: Non-Inferiority — Non-inferiority of AdreView™ group over SoC group was demonstrated if upper bound of the 95% confidence interval (CI) for the hazard ratio (HR) (AdreView™ group / SoC) was equal to 1.20; p = 0.8459, Log Rank — Threshold for significance at 0.025 level; Hazard Ratio (HR) = 1.047, 95% CI 2-sided [0.295 to 3.719] — AdreView™ vs. Standard of Care

2. Secondary Outcome: Percentage of Participants With Events of Complications of Device: H/M >=1.6 in Full Analysis Set
Description: Composite of the percentage of participants with events of hospitalization or death related to major complications of device implantation (i.e., need for thoracotomy, pericardiocentesis, or vascular surgery), complications of long-term device therapy (i.e., infection not leading to hospitalization, lead and/or generator removal/replacement, inappropriate shocks, explanation), and combined as 'complications of device' for participants with H/M >=1.6. Participants who were alive at time of database lock (DBL) were censored at the last known-alive date.
Time Frame: From randomization until the end of the follow-up period (median 304 days)
Population: Analysis was performed on FAS population. Here, overall number of participants analyzed = participants with H/M >=1.6.
Measure: Number; unit: percentage of participants
Arm/Group | AdreView™ | Standard of Care
Number analyzed (Participants) | 26 | 20
percentage of participants
  Hospitalization/death | 3.8 | 0
  Complications of long-term device therapy | 3.8 | 15.0
  Complications of device | 3.8 | 15.0

3. Secondary Outcome: Percentage of Participants With Cardiac Death
Description: Cardiac death composed of sudden cardiac death, death due to cardiac arrhythmia, death due to heart failure, and death due to other cardiovascular causes.
Time Frame: From randomization until the end of the follow-up period (median 304 days)
Population: Analysis was performed on FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | AdreView™ | Standard of Care
Number analyzed (Participants) | 164 | 157
percentage of participants | 1.2 | 0.6

4. Secondary Outcome: Percentage of Participants With Hospitalization for Cardiovascular Cause
Description: Percentage of participants who were hospitalized for cardiovascular cause were reported.
Time Frame: From randomization until the end of the follow-up period (median 304 days)
Population: Analysis was performed on FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | AdreView™ | Standard of Care
Number analyzed (Participants) | 164 | 157
percentage of participants | 7.3 | 7.6

5. Secondary Outcome: Percentage of Participants With All-Cause Hospitalization
Description: Percentage of participants with all-cause hospitalization were reported.
Time Frame: From randomization until the end of the follow-up period (median 304 days)
Population: Analysis was performed on FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | AdreView™ | Standard of Care
Number analyzed (Participants) | 164 | 157
percentage of participants | 17.1 | 22.3

6. Secondary Outcome: Percentage of Participants With Events (Composite of the Occurrence of Resuscitated Life-Threatening Ventricular Tachycardia, Unstable Ventricular Tachyarrhythmias, Sudden Cardiac Death [SCD] and Resuscitated Cardiac Arrest)
Description: Percentage of participants with composite events i.e occurrence of resuscitated life-threatening ventricular tachycardia, unstable ventricular tachy-arrhythmias, SCD and resuscitated cardiac arrest were reported. Participants who were alive at time of database lock (DBL) were censored at the last known-alive date.
Time Frame: From randomization until the end of the follow-up period (median 304 days)
Population: Analysis was performed on FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | AdreView™ | Standard of Care
Number analyzed (Participants) | 164 | 157
percentage of participants | 1.2 | 2.5

7. Secondary Outcome: Percentage of Participants With Syncope
Description: Percentage of participants with Syncope were reported. Participants who were alive at time of DBL were censored at the last known-alive date by date of DBL.
Time Frame: From randomization until the end of the follow-up period (median 304 days)
Population: Analysis was performed on FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | AdreView™ | Standard of Care
Number analyzed (Participants) | 164 | 157
percentage of participants | 2.4 | 0

8. Secondary Outcome: Percentage of Participants With Implantable Cardioverter Defibrillator (ICD) Implantation
Description: Percentage of participants with ICD implantation were reported.
Time Frame: From randomization until the end of the follow-up period (median 304 days)
Population: Analysis was performed on FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | AdreView™ | Standard of Care
Number analyzed (Participants) | 164 | 157
percentage of participants | 73.2 | 81.5

9. Secondary Outcome: Percentage of Participants With Events of Complications of Device
Description: Composite of the percentage of participants with events of hospitalization or death related to major complications of device implantation (i.e., need for thoracotomy, pericardiocentesis, or vascular surgery), complications of long-term device therapy (i.e., infection not leading to hospitalization, lead and/or generator removal/replacement, inappropriate shocks, explanation), and combined as 'complications of device'.
Time Frame: From randomization until the end of the follow-up period (median 304 days)
Population: Analysis was performed on FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | AdreView™ | Standard of Care
Number analyzed (Participants) | 164 | 157
percentage of participants
  Hospitalization/death | 4.9 | 3.8
  Complications of long-term device therapy | 4.3 | 6.4
  Complications of device | 5.5 | 6.4

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from randomization until the end of the follow-up period (median 304 days) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are study-emergent AEs that is AEs and deaths that developed/worsened during any time after randomization until end of the follow-up period (median 304 days). Analysis was performed on safety population which included all participants who signed the informed consent form and met all the inclusion criteria and none of the exclusion criteria.
Groups:
- Total Participants: All participants who were randomized in AdreView™ and Standard of Care group in addition with non-randomized participants who signed informed consent form.
Arm/Group | AdreView™ | Standard of Care | Total Participants
All-Cause Mortality (participants affected / at risk) | 6/164 | 5/157 | 11/343
Serious Adverse Events (participants affected / at risk) | 65/164 | 62/157 | 127/343
Other Adverse Events (participants affected / at risk) | 0/164 | 0/157 | 0/343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AdreView™ (N=164) | Standard of Care (N=157) | Total Participants (N=343)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 2 | 3
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 5 | 2 | 7
Atrial fibrillation (Cardiac disorders) | 3 | 3 | 6
Cardiac arrest (Cardiac disorders) | 3 | 1 | 4
Cardiac disorder (Cardiac disorders) | 26 | 22 | 48
Cardiac failure (Cardiac disorders) | 8 | 5 | 13
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 3
Cardiac perforation (Cardiac disorders) | 2 | 0 | 2
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 2
Tachycardia (Cardiac disorders) | 0 | 2 | 2
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 2 | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 1 | 4 | 5
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Chest discomfort (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 1
Complication associated with device (General disorders) | 1 | 1 | 2
Malaise (General disorders) | 1 | 0 | 1
Medical device site irritation (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 2
Pain (General disorders) | 1 | 0 | 1
Polyp (General disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 0 | 3
Cellulitis (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 1
Gangrene (Infections and infestations) | 0 | 1 | 1
Helicobacter infection (Infections and infestations) | 0 | 1 | 1
Implant site infection (Infections and infestations) | 0 | 1 | 1
Incision site infection (Infections and infestations) | 1 | 0 | 1
Infection (Infections and infestations) | 1 | 1 | 2
Influenza (Infections and infestations) | 2 | 3 | 5
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2
Otitis media (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1 | 5
Post procedural cellulitis (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Sepsis (Infections and infestations) | 2 | 0 | 2
Septic shock (Infections and infestations) | 0 | 1 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Viral infection (Infections and infestations) | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1
Blood uric acid increased (Investigations) | 2 | 0 | 2
C-reactive protein increased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastrointestinal stro (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 2
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 4 | 1 | 5
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Device inappropriate shock delivery (Product Issues) | 3 | 2 | 5
Device use issue (Product Issues) | 1 | 1 | 2
Lead dislodgement (Product Issues) | 2 | 2 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 3
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 2 | 1 | 3
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1 | 1
Circulatory collapse (Vascular disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 2 | 1 | 3
Intermittent claudication (Vascular disorders) | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was early terminated by sponsor after enrollment of 395 participants due to very slow recruitment rates. Sample size was 395 participants instead of planned 2354 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.

DOCUMENTS (2):
  • Study Protocol (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT02656329/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT02656329/SAP_001.pdf